CLINICAL TRIAL: NCT06034444
Title: Better tArgetting, Better Outcomes for Frail ELderly Patients: A Quality Improvement Initiative in Long-term Care Facilities Using interRAI Long-term Care Assessment in Quebec
Brief Title: Better tArgetting, Better Outcomes for Frail ELderly Patients
Acronym: BABEL
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Sponsor
Other Study IDs: 17.205
Record Dates: First submitted 2018-06-20; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Residents in Longterm Care Facilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- interRAI LTCF: Nursing homes in Quebec where interRAI evaluations and care plans will be introduced.
  Interventions: Other: interRAI LTCF

INTERVENTIONS:
Other: interRAI LTCF — Standardized evaluations (interRAI LTCF) will be introduced to selected nursing homes in Quebec.

SUMMARY:
The acronym for this proposal, BABEL, refers to the fact that a common "language" - the interRAI risk-stratification and decision-making tool - will be used in this project, allowing several measures of care quality in long-term care facilities to be compared with those in other provinces for the first time. The impact of the use of this assessment system and associated care planning protocols will also be investigated using usual practice as the point of reference.

ELIGIBILITY:
Inclusion Criteria:

* All nursing home residents in a particular unit where standardized evaluations are being introduced (for example, all residents in a particular floor or wing of the longterm care facility)

Exclusion Criteria:

* Residents who are admitted to a nursing home unit for less than 1 week.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents in a long-term care facility (nursing home)
Sampling Method: Non-Probability Sample
Enrollment: 5692 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in depression prevalence | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  Depression rating scale score of 3 or more (from interRAI LTCF)
Change in prevalence of potentially inappropriate antipsychotic use | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  Use of antipsychotics in the absence of an appropriate diagnosis
Change in falls prevalence | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  Prevalence of falls among residents under study
Change in prevalence of pain | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  Using interRAI pain scale scores greater than 0
Change in the prevalence of physical restraints use | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  Use of physical restraints on residents as assessed using interRAI LTCF

SECONDARY OUTCOMES:
Change in prevalence of pressure ulcers | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  Stage 2 pressure ulcer on the interRAI pressure ulcer scale

OTHER OUTCOMES:
Change in other interRAI LTCF quality indicators | Every 3 months, for a minimum of 6 months and a maximum of 36 months
  interRAI LTCF evaluation leads to a number of quality indicators being generated each of which will be tracked over time for each facility to compare before and after effects, as well as comparisons with other centers in Canada

CONTACTS AND LOCATIONS:
Locations (1):
- Donald Berman Maimonides, Montreal, Quebec, Canada